CLINICAL TRIAL: NCT07249424
Title: Evaluation of the Effective Myocardial Protection Duration of Del Nido Cardioplegia: A Prospective Observational Study in Adult Patients Undergoing Cardiac Surgery
Brief Title: Effective Myocardial Protection Time of Del Nido Cardioplegia in Adult Cardiac Surgery
Acronym: DN-TIME-2025
Status: Recruiting | Type: Observational
Sponsor: Muhammet Talha Ceran, MD (Other)
Responsible Party: Sponsor-Investigator, Muhammet Talha Ceran, MD, Cardiovascular Surgery Resident, Principal Investigator, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Other Study IDs: E-40209705-050.01-1123786
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Heart Valve Diseases; Aortic Diseases; Myocardial Ischemia; Reperfusion Injury, Myocardial; Postoperative Complications (Cardiopulmonary); Cardiopulmonary Bypass
Keywords: Del Nido cardioplegia; cardioplegia; aortic cross-clamp (ACC); high-sensitivity troponin; myocardial protection; cardiopulmonary bypass (CPB); aortic cross-clamp time; single-dose cardioplegia; ischemia-reperfusion; valve surgery; thoracic aortic surgery
MeSH Terms: conditions — Heart Valve Diseases; Aortic Diseases; Myocardial Ischemia; Myocardial Reperfusion Injury; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Del Nido Cardioplegia Cohort: Adults undergoing elective valve and/or thoracic aortic surgery under CPB with ACC in which Del Nido cardioplegia is used per routine practice. No experimental therapy; only study-specific blood sampling for hs-troponin at predefined times.

SUMMARY:
This single-center, prospective, observational cohort study quantifies the effective myocardial protection window of Del Nido cardioplegia during adult open-heart surgery performed under cardiopulmonary bypass (CPB) and aortic cross-clamp (ACC). Without altering routine care, time-stamped high-sensitivity cardiac troponin (hs-cTn) measurements will be obtained at predefined intraoperative and early postoperative intervals to identify the inflection ("change-point") at which biochemical evidence of ischemic injury begins to rise. Eighty adults undergoing elective valve and/or thoracic aortic procedures with Del Nido cardioplegia will be enrolled. The primary endpoint is the intraoperative hs-cTn change-point time referenced to ACC. Secondary endpoints include associations between change-point and ACC duration, the presence/timing of any re-dose, and early clinical outcomes (e.g., low cardiac output syndrome, maximum VIS in the first 24 h, new arrhythmia or pacemaker need, acute kidney injury by KDIGO, ventilation hours, ICU/hospital length of stay, 30-day MACE and mortality). All cardioplegia choices (dose, route, temperature, re-dose decisions) remain per standard practice; no experimental therapy is administered. Risks are minimal and limited to small-volume blood sampling coordinated with routine draws.

DETAILED DESCRIPTION:
Background and Rationale Del Nido cardioplegia is widely used in adult valve/aortic surgery to permit prolonged single-dose electrical arrest. The effective protection duration likely varies with patient and procedural factors (e.g., LV function, temperature, hemodilution, surgical complexity, antegrade/retrograde delivery). Many centers empirically re-dose around 60-90 minutes; however, this window may not be optimal for every case. The current study quantifies the protection window by coupling routine care with dense, time-stamped hs-troponin sampling.

Design and Setting Prospective, single-center, observational cohort conducted at Necmettin Erbakan University, Department of Cardiovascular Surgery (Türkiye).

Population Adults 18-80 years scheduled for elective valve and/or thoracic aortic surgery under CPB with ACC in which Del Nido cardioplegia is used per institutional routine. Key exclusions include isolated or CABG-dominant procedures, redo sternotomy, emergency/salvage or preoperative shock, IABP/ECMO, LVEF <35%, eGFR <45 mL/min/1.73 m², significant pulmonary or hepatic disease, major coagulopathy, active infection/sepsis or endocarditis, pregnancy, and preoperative troponin elevation.

Interventions None. Cardioplegia content, dose, route (antegrade/retrograde/combined), temperature, and re-dose decisions are entirely per standard practice at the discretion of the surgical/anesthesia/perfusion team. No experimental therapy is administered.

Sampling Schedule (Biomarkers) Preoperative baseline hs-cTn; intraoperative sampling referenced to ACC at 0, 30, and 60 minutes, then intensified at 75, 90, 105, and 120 minutes. If a re-dose is administered, additional samples at pre-re-dose and +15/+30/+45/+60 minutes. Postoperative hs-cTn at approximately 6, 24, and 48 hours. Intraoperative blood is obtained preferably from the venous reservoir or existing central lines. Each draw ~3-5 mL; total additional volume ~30-40 mL. Exploratory CK-MB may be recorded where available.

Outcomes Primary outcome: intraoperative hs-cTn change-point time (minutes from ACC) identified by segmented (piecewise) trend analysis indicating the earliest sustained acceleration compatible with evolving ischemic injury.

Key secondary outcomes: (i) association between change-point and ACC duration; (ii) presence/timing of Del Nido re-dose and biochemical response to re-dose (slope change pre/post); (iii) early clinical outcomes including low cardiac output syndrome, maximum VIS in the first 24 h, new arrhythmia or pacemaker need, acute kidney injury by KDIGO, ventilation hours, ICU/hospital length of stay, re-exploration/bleeding, infection, 30-day MACE, and 30-day all-cause mortality.

Statistical Plan (Summary) Individual time series will be analyzed using segmented (piecewise) regression and/or change-point detection methods. Group-level estimates (mean protection window and variance) will be obtained via mixed-effects change-point models. Associations with durations (ACC, CPB), re-dose timing, and outcomes will use linear/quantile regression and logistic/Poisson/negative binomial models as appropriate. Missing data will be handled per predefined rules and, if needed, multiple imputation. Target enrollment is 80 participants, anticipated to provide ~80% power at α=0.05 to detect a clinically meaningful change-point and slope shift in hs-troponin trajectories.

Safety and Data Handling Risk is minimal and limited to low-volume blood sampling aligned with routine care; no experimental treatment is given. Data are recorded on standardized case report forms and stored in secure, de-identified systems compliant with local regulations. Serious adverse events are reported per institutional/authority requirements.

Significance By quantifying the actual protection window and its variability, the study is designed to inform more rational-potentially individualized-re-dose timing for Del Nido cardioplegia, aiming to reduce both under-protection (late re-dose) and workflow disruption (unnecessary early re-dose).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Elective valve surgery (aortic, mitral, tricuspid), thoracic aortic surgery, or combined valve + thoracic aortic procedures
* Planned cardiopulmonary bypass (CPB) with aortic cross-clamp (ACC)
* Use of Del Nido cardioplegia per institutional routine
* Ability to provide written informed consent (participant or legally authorized representative)

Exclusion Criteria:

* Isolated CABG or CABG-dominant combined procedures
* Redo sternotomy
* Emergency status (including shock) or preoperative mechanical circulatory support (IABP or ECMO), or anticipated need for such support
* Left ventricular ejection fraction <35%
* Estimated GFR <45 mL/min/1.73 m²
* Moderate-severe chronic lung disease with significant functional limitation, or severe pulmonary hypertension
* Active infection/sepsis or active infective endocarditis
* Severe hepatic dysfunction, major coagulopathy, or bleeding diathesis
* Pregnancy
* Deep hypothermia protocols (<28 °C)
* Procedures without ACC
* Preoperative cardiac troponin above the laboratory upper reference limit
* Any condition that, in the judgment of the treating team, would preclude safe participation or protocol adherence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single-center, tertiary academic cardiovascular surgery service at Necmettin Erbakan University Meram Medical Faculty Hospital (Konya, Türkiye). Consecutive adults (18-80 years) undergoing elective valve and/or thoracic aortic surgery with cardiopulmonary bypass and aortic cross-clamping, in whom Del Nido cardioplegia is used as part of routine care, are screened and, if eligible, approached for written informed consent. Approximately 80 participants are enrolled and followed through the index hospitalization; 30-day outcomes are abstracted from the medical record/standard follow-up. Observational cohort; no randomization; all treatment decisions per usual care.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hs-troponin change-point time (minutes from ACC) | From aortic cross-clamp (ACC) application to 120 minutes intraoperatively; if a re-dose is given, up to 60 minutes after the re-dose within the same operation.
  For each participant, serial hs-cTn values obtained at ACC 0/30/60/75/90/105/120 minutes (and at re-dose pre/+15/+30/+45/+60 when applicable) will be modeled with segmented (piecewise) regression. The change-point is defined as the earliest time with a statistically significant increase in slope indicating evolving myocardial injury. Unit: minutes; lower values reflect earlier loss of protection.

SECONDARY OUTCOMES:
Biochemical response to re-dose (slope change in hs-troponin) | From re-dose (time 0) to +60 minutes intraoperatively.
  Within-subject comparison of hs-cTn trajectory slope before vs after re-dose using segmented regression. Metric: difference in slopes (ng/L per minute).
Peak postoperative hs-troponin (0-48 h) | From end of surgery to 48 hours postoperatively (samples ~6, 24, 48 h).
  Maximum measured hs-cTn (ng/L) within the first 48 hours after surgery.
Low Cardiac Output Syndrome (LCOS) within 24 hours | First 24 postoperative hours.
  LCOS defined as any of the following: (a) maximum vasoactive-inotropic score (VIS) ≥15 for ≥2 consecutive hours; or (b) initiation of mechanical circulatory support (IABP/ECMO); or (c) cardiac index <2.2 L/min/m² with clinical hypoperfusion requiring inotrope/vasopressor escalation. Outcome reported as proportion of participants meeting criteria.
30-day major adverse cardiovascular events (MACE) | 30 days after surgery
  Composite of all-cause death, non-fatal myocardial infarction (per institutional cardiac-surgery definition), and stroke/TIA. Reported as proportion of participants; components also summarized separately.

OTHER OUTCOMES:
Association between change-point time and ACC duration | Intraoperative (from ACC on to 120 min; re-dose window as applicable)
  Linear/quantile regression of change-point time (min) on ACC duration (min). Effect size reported as β per 10-min increase in ACC with 95% CI.
Immediate reperfusion arrhythmia after ACC removal | From ACC removal to 30 minutes after reperfusion
  Incidence of VF/VT requiring defibrillation or temporary pacing. Reported as proportion; association with change-point explored.

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Dereli, Prof. Dr., Principal Investigator — Necmettin Erbakan University, Dept. of Cardiovascular Surgery; Muhammet Talha Ceran, Principal Investigator — Necmettin Erbakan University, Dept. of Cardiovascular Surgery
Locations (1):
- Necmettin Erbakan University Meram Faculty of Medicine, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the primary and key secondary outcomes (time-stamped hs-troponin values, basic demographics, operative variables, and early postoperative outcomes). Data will be shared in compliance with local regulations (e.g., KVKK) and institutional policies.
Supporting Information: Study Protocol, SAP
Time Frame: Available beginning 6-12 months after the primary publication (or within 12 months after last-patient-last-visit if no publication) and will remain available for 5 years.
Access Criteria: Qualified researchers may request access by submitting a brief proposal to the Central Contact. Requests will be reviewed by the study investigators and the institutional Data Access Committee. Upon approval and execution of a Data Use Agreement (non-reidentification, secure storage, academic use only, citation/acknowledgment, and data destruction at project end), de-identified IPD and supporting documents will be transferred via secure link.
  Central Contact: Muhammet Talha Ceran, MD - mtceran@gmail.com
URL: https://hastane.erbakan.edu.tr

REFERENCES:
- [Result] Devereaux PJ, Lamy A, Chan MTV, Allard RV, Lomivorotov VV, Landoni G, Zheng H, Paparella D, McGillion MH, Belley-Cote EP, Parlow JL, Underwood MJ, Wang CY, Dvirnik N, Abubakirov M, Fominskiy E, Choi S, Fremes S, Monaco F, Urrutia G, Maestre M, Hajjar LA, Hillis GS, Mills NL, Margari V, Mills JD, Billing JS, Methangkool E, Polanczyk CA, Sant'Anna R, Shukevich D, Conen D, Kavsak PA, McQueen MJ, Brady K, Spence J, Le Manach Y, Mian R, Lee SF, Bangdiwala SI, Hussain S, Borges FK, Pettit S, Vincent J, Guyatt GH, Yusuf S, Alpert JS, White HD, Whitlock RP; VISION Cardiac Surgery Investigators. High-Sensitivity Troponin I after Cardiac Surgery and 30-Day Mortality. N Engl J Med. 2022 Mar 3;386(9):827-836. doi: 10.1056/NEJMoa2000803. PMID 35235725
- [Result] Behrendt T. Scanning densitometer for photographic fundus measurements. Am J Ophthalmol. 1966 Oct;62(4):689-93. doi: 10.1016/0002-9394(66)92195-7. No abstract available. PMID 5929134
- [Result] McGrath S, Alaour B, Kampourakis T, Marber M. Cardiac Troponin: Fragments of the Future? JACC Adv. 2025 May;4(5):101695. doi: 10.1016/j.jacadv.2025.101695. Epub 2025 Apr 25. PMID 40286361
- [Result] Nakao M, Morita K, Shinohara G, Kunihara T. Modified Del Nido Cardioplegia and Its Evaluation in a Piglet Model. Semin Thorac Cardiovasc Surg. 2021 Spring;33(1):84-92. doi: 10.1053/j.semtcvs.2020.03.002. Epub 2020 May 7. PMID 32387781
- [Result] Januzzi JL Jr. Troponin testing after cardiac surgery. HSR Proc Intensive Care Cardiovasc Anesth. 2009;1(3):22-32. PMID 23439987
- [Result] Eris C, Engin M, Erdolu B, Kagan As A. Comparison of del Nido Cardioplegia vs. blood cardioplegia in adult aortic surgery: Is the single-dose cardioplegia technique really advantageous? Asian J Surg. 2022 May;45(5):1122-1127. doi: 10.1016/j.asjsur.2021.09.032. Epub 2021 Oct 12. PMID 34649799